CLINICAL TRIAL: NCT02323399
Title: Phase 4 Open Label Study to Determine Pharmacokinetics of Phenylephrine and Pharmacodynamic Effects on BP Via IV Admin of Phenylephrine Hydrochloride Inj in Ped Subjects (≥12 to 16 Years of Age) Undergoing Gen and Neuraxial Anesthesia
Brief Title: Study to Determine the Pharmacokinetics and Pharmacodynamic Effects of Phenylephrine on BP Via IV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: West-Ward Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1420RDP009
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phenylephrine (Experimental): Phenylephrine Hydrochloride Injection, USP (United States Pharmacopeia) 10 mg/mL label claim
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine — one of six initial treatments Phenylephrine Hydrochloride Injection (PHI) will be initially administered to approximately 50 subjects as an intravenous bolus (IV-B) at Low (1 μg/kg), Med (3 μg/kg), or High (5 μg/kg) level; PHI will be initially administered to approximately 50 subjects as a continuous intravenous infusion (IV-I) at Low (0.25 μg/kg/min), Med (0.75 μg/kg/min), or High (1.25 μg/kg/min) level]; each initial treatment group will have two PK sampling schedules.
  Other Names: Phenylephrine Hydrochloride Injection

SUMMARY:
The primary objective of this study is to evaluate the dose effect of Phenylephrine Hydrochloride Injection on the treatment of clinically relevant decreased blood pressure in the pediatric population, ≥12 to 16 year old patients undergoing general and neuraxial anesthesia.

The secondary objectives are to describe changes in blood pressure and heart rate, time to onset and to maximal response, and the duration of response; to assess the safety of the product in this population; and to characterize the pharmacokinetics of phenylephrine hydrochloride.

DETAILED DESCRIPTION:
This is a Phase 4 multi-center, randomized open-label study in 100 subjects aged ≥12 to 16 years who experience a decrease in blood pressure during a procedure requiring general or neuraxial anesthesia. At least 300 subjects will be enrolled in this study. It is anticipated that up to 33% of enrolled subjects will actually experience a decrease in blood pressure that requires treatment and so will receive Phenylephrine Hydrochloride Injection (PHI). There are 12 possible randomization assignments: one of six initial treatments PHI will be initially administered to approximately 50 subjects as an intravenous bolus (IV-B) at Low (1 μg/kg), Med (3 μg/kg), or High (5 μg/kg) level; PHI will be initially administered to approximately 50 subjects as a continuous intravenous infusion (IV-I) at Low (0.25 μg/kg/min), Med (0.75 μg/kg/min), or High (1.25 μg/kg/min) level]; each initial treatment group will have two pharmacokinetics (PK) sampling schedules.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age is between ≥12 and 16 years, inclusive
2. Subject is scheduled for a procedure that requires general or neuraxial anesthesia
3. Subjects must have normal or clinically acceptable physical exam
4. Subjects with controlled diabetes prior to entry must have a mean systolic/diastolic office blood pressure ≤128/78 mmHg (sitting, after 5 minutes of rest)
5. Females must have a urine or serum pregnancy test (Human Chorionic Gonadotropin) that is negative at Screening and Day 1
6. Subject's parent or legal guardian gives informed consent and subject gives assent.

Exclusion Criteria:

1. Subject has a contraindication to vasoconstrictor therapy for control of blood pressure
2. Subject has participated in other clinical trials for investigational drugs and/or devices within 30 days prior to enrollment
3. Subject has any serious medical condition which, in the opinion of the investigator, is likely to interfere with study procedures
4. Subjects who have a history of any clinically significant local or systemic infectious disease within four weeks prior to initial treatment administration
5. Subjects who are positive for hepatitis B surface antigen or hepatitis C antibody
6. Subjects taking antihypertensive medication
7. Subject is moribund (death is likely to occur in less than 48 hours)
8. Females who are pregnant, nursing or unwilling to use/practice adequate contraception.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Plasma Phenylephrine (PE) concentrations will be measured using a validated liquid chromatography/mass spectrometry (LCMS/MS) assay. | Screening up to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Ormeno, MD, Study Director — PRA Health Sciences
Locations (10):
- United States (10):
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Jackson Memorial Hospital, Miami, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Stony Brook Medicine, Stony Brook, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Medical Center of Dallas, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Ruby Memorial Hospital, Morgantown, West Virginia